CLINICAL TRIAL: NCT01644929
Title: Rehabilitation Combined With Bihemispherictranscranial Direct Current Stimulation in Subacute Ischemic Stroke to Increase Upper Limb Motor Recovery, a Randomised, Controlled, Double-blind Study
Brief Title: Rehabilitation Combined With Bihemispherictranscranial Direct Current Stimulation in Subacute Ischemic Stroke
Acronym: RECOMBINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. med. Carlo Cereda (Other Government)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Clinica Hildebrand Brissago (Other); Advisory Board Research Ente Ospedaliero Cantonale (Unknown)
Responsible Party: Sponsor-Investigator, Dr. med. Carlo Cereda, Capo clinica, Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EOC.NSI.11.02
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: First Ever Clinical Stroke; Ischemic Stroke; Subacute Phase; Persistent Hemiparesis of Upper Extremity
Keywords: hemiparesis; bihemispheric transcranial direct current stimulation; ischemic stroke; subacute; rehabilitation; physiotherapy; ergotherapy
MeSH Terms: conditions — Ischemic Stroke; Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 tDCS-Sham (Experimental): tDC stimulation for 3 weeks, then cross-over to sham stimulation
  Interventions: Procedure: transcranial direct current stimulation (tDCS)
- 2 Sham-tDCS (Experimental): Sham stimulation for 3 weeks, then cross over to tDCS stimulation
  Interventions: Procedure: Sham stimulation, then tDCS
- 3 Sham-Sham (Sham Comparator): Treatment for 6 weeks daily with sham stimulation
  Interventions: Procedure: Sham stimulation

INTERVENTIONS:
Procedure: transcranial direct current stimulation (tDCS) — Anodal tDCS of the ipsilesional motor cortex and cathodal tDCS of contralesional motor cortex (1.5 mA, 30 minutes) for 15 days during three weeks, then sham stimulation for 30 seconds on 15 days during 3 weeks
  Arms: 1 tDCS-Sham
Procedure: Sham stimulation, then tDCS — Sham stimulation for 30 seconds on 15 days during 3 weeks, then anodal tDCS of the ipsilesional motor cortex and cathodal tDCS of contralesional motor cortex (1.5 mA, 30 minutes) for 15 days during three weeks
  Arms: 2 Sham-tDCS
Procedure: Sham stimulation — Sham stimulation for 30 seconds on 15 days during 6 weeks
  Arms: 3 Sham-Sham

SUMMARY:
Rehabilitation after stroke improves motor functions by promoting plastic changes however, after completing standard rehabilitation, 50-60% of patients still exhibit some degree of motor impairment and require at least partial assistance in activities of day living. Therefore, the exploration of other approaches to promote recovery is compulsory. Non invasive brain stimulation and motor rehabilitation are thought to share similar mechanisms in inducing neuroplastic changes in the human cortex and an emerging field of research is focusing on the possibility of coupling both therapies in order to achieve an additive effect and improve outcome.

We hypothesize that coupling bihemispheric transcranial direct current stimulation (tDCS) with simultaneous physical/occupational therapy in the subacute phase of ischemic stroke patients may improve upper limb motor recovery in humans.

This is a randomized, controlled, double blind, cross-over, multicentre, clinical trial. Thirty-six ischemic stroke patients in the subacute phase will be recruited in three centers of neurorehabilitation in Switzerland. After stratification based on the Fugl-Meyer Assessment Upper Extremity according to the severity of the deficit, the patient will be randomized to receive besides standardized physical/occupational treatment according to the Impairment-Oriented Training, tDCS of themotor cortex (1.5 mA, 30 minutes) (group 1: 12 patients) or sham stimulation (without current) (group 2: 12 patients). After three weeks of treatment group 1 and 2 will cross-over and will be treated for other three weeks. Group 3 (12 patients) will receive routine physical/occupational treatment and sham tDCS for six weeks. Assessment will be performed before starting tDCS, at week 3, 6 and at 6 months. Outcome measures are the Fugl-Meyer Assessment Upper Extremity, the extended Barthel Index, the Ashworth scale, the Test of Upper Limb Apraxia (only baseline, week 6, month6), the grip strength evaluated by the Jamar Hydraulic Hand dynamometer. At baseline at week 6 and at month 6 depression will be assessed by the Hamilton depression Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic lesions in the territory of middle cerebral artery subcortical or subcortical/cortical confirmed neuroimaging
2. Inclusion must be in the sub-acute phase defined as within 2-4 weeks after stroke
3. Persistent hemiparesis, indicated by a score of 1-3 on the motor arm item of the NIH Stroke Scale (NIHSS) (Brott et al. 1989) but wrist and finger movement is not required
4. No UE injury or conditions that limited use prior to the stroke.
5. The patient is >18 years old.
6. The patient has subscribed the informed consent

Exclusion Criteria:

1. History of epilepsy, brain tumor, major head trauma, learning disorder, severe cognitive impairment, drug or alcohol abuse, major psychiatric illness
2. Use of medications that may lower seizure threshold (e.g., metronidazole, fluoroquinolones)
3. Severe pain in the affected upper limb (>=8 on the shoulder item of the "joint pain during passive motion" of the Fugl-Meyer Assessment Upper Extremity)
4. Further stroke or other significant medical complication during the study
5. Evidence of severe leucoencephalopathy (grade IV according to the Fazeka's scale)
6. Important aphasia that would impair the understanding and performance of the assessment scales

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity | 6 weeks
  Investigator administered questionnaire

SECONDARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity | 3 weeks
  Investigator administered questionnaire
Fugl-Meyer Assessment Upper Extremity | 6 months
  Investigator administered questionnaire
Barthel Index | 3 weeks
  Investigator administered questionnaire
Barthel Index | 6 weeks
  Investigator administered questionnaire
Barthel Index | 6 months
  Investigator administered questionnaire
Ashworth scale | 3 weeks
  Investigator administered questionnaire
Ashworth scale | 6 weeks
  Investigator administered questionnaire
Ashworth scale | 6 months
  Investigator administered questionnaire
Test of Upper Limb Apraxia (TULIA) | 6 weeks
  investigator administered questionnaire
Test of Upper Limb Apraxia (TULIA) | 6 months
  investigator administered questionnaire
Grip strength | 3 weeks
  Jamar Hydraulic Hand dynamometer
Grip strength | 6 weeks
  Jamar Hydraulic Hand dynamometer
Grip strength | 6 months
  Jamar Hydraulic Hand dynamometer
Hamilton depression Rating scale | 6 weeks
  Patient administered questionnaire
Hamilton depression Rating scale | 6 months
  Patient administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Cereda, MD, Principal Investigator — Ospedale Regionale di Lugano - Civico
Locations (3):
- Switzerland (3):
  - Universitätsspital Bern, Inselspital, Neuropsychologische Rehabilitation, Bern
  - Clinica Hildebrand, Centro di riabilitazione Brissago, Brissago
  - HELIOS Klinik Zihlschlacht AG, Neurologisches Rehabilitationszentrum, Zihlschlacht

REFERENCES:
- [Background] Lindenberg R, Renga V, Zhu LL, Nair D, Schlaug G. Bihemispheric brain stimulation facilitates motor recovery in chronic stroke patients. Neurology. 2010 Dec 14;75(24):2176-84. doi: 10.1212/WNL.0b013e318202013a. Epub 2010 Nov 10. PMID 21068427
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- See also: Link to the hospital coordinating the study — http://www.eoc.ch
- See also: Link to the hospital participating in the study — http://neurologie.insel.ch/de/
- See also: Link to the clinic participating in the study — http://www.clinica-hildebrand.ch/